CLINICAL TRIAL: NCT05672862
Title: International Post-PCI FFR Registry for Extended Follow up Outcomes After Coronary Stenting
Brief Title: International Post-PCI FFR Extended Registry
Status: Completed | Type: Observational
Sponsor: Bon-Kwon Koo (Other)
Collaborators: Inje University Ilsan Paik Hospital, Goyang, South Korea (Unknown); Nanjing First Hospital, Nanjing Medical University, Nanjing, China (Unknown); Tsuchiura Kyodo General Hospital (Other); Gifu Heart Center, Gifu, Japan (Unknown); Keimyung University Dongsan Medical Center, Daegu, South Korea (Unknown); Ulsan University Hospital, Ulsan, South Korea (Unknown); Samsung Medical Center (Other); Kyoto Second Red Cross Hospital, Kyoto, Japan (Unknown); Sejong General Hospital (Other)
Responsible Party: Sponsor-Investigator, Bon-Kwon Koo, Professor, Seoul National University Hospital
Organization: Seoul National University Hospital (Other)
Other Study IDs: H-2108-211-1251
Record Dates: First submitted 2021-11-04; First posted 2023-01-05 (Actual); Last update posted 2023-01-31 (Actual); Status verified 2023-01

CONDITIONS: Coronary Disease
Keywords: fractional flow reserve; percutaneous coronary intervention; drug-eluting stent; coronary atherosclerosis
MeSH Terms: conditions — Coronary Disease; Coronary Artery Disease | interventions — Percutaneous Coronary Intervention

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Post PCI state: The study population of this study underwent percutaneous coronary intervention(PCI) with drug-eluting stent (DES) and measured fractional flow reserve after PCI.
  Interventions: Device: Percutaneous coronary intervention

INTERVENTIONS:
Device: Percutaneous coronary intervention — PCI was performed using drug-eluting stents

SUMMARY:
Percutaneous coronary intervention (PCI) is a standard treatment strategy for coronary artery disease (CAD). With the presence of myocardial ischemia, PCI reduces the risks of death, myocardial infarction (MI), and revascularization compared to medical therapy. However, the risk of future clinical events remains high, and about 10% of patients experienced further cardiovascular events after PCI. Several factors are associated with these poor outcomes. Well-known patient-related risk factors are diabetes mellitus, chronic kidney disease, left ventricular dysfunction, previous MI, and presentation with acute coronary syndrome. Procedure-related factors, such as stent under expansion, malposition, edge dissection, the number of the used stent, and total stent length, are also related to poor prognosis after PCI. Recent studies reported that fractional flow reserve (FFR) after coronary stenting, or post-PCI FFR, was associated with future clinical outcomes after PCI, and low post-PCI FFR value was associated with procedural factors. However, optimal cut-off values of post-PCI FFR ranged widely, from 0.86 to 0.96, and some studies reported the limited prognostic value of post-PCI FFR. This might result from differences in study populations, the definition of outcomes, type of stent used, and distribution of included vessels among previous studies. Previously, the investigators incorporated previous data into the International Post-PCI FFR registry and demonstrated the prognostic value of post-PCI FFR using the machine learning technique. However, the results were based on the two years follow-up of patients after PCI, and the prognostic value of post-PCI FFR in long-term outcomes is still uncertain. Therefore, the investigators planned to extend the International Post-PCI FFR registry to define the long-term prognostic implication of post-PCI FFR.

DETAILED DESCRIPTION:
The investigators planned to extend the International Post-PCI FFR registry (NCT04684043) to explore the long-term prognostic value of post-PCI FFR. The International Post-PCI FFR registry (NCT04684043) already included the 2,200 patients who underwent PCI and measured post-PCI FFR between June 2011 and May 2018. As the clinical, angiographic, and physiologic data are already collected in the International Post PCI FFR registry, the investigators will further collect the most recent clinical outcome data until 2021.5 and incorporate them into the International Post-PCI FFR Extended registry. As the current study will evaluate clinical outcomes at 5 years, 2,128 patients who underwent PCI and measured post-PCI FFR between June 2011 and Nov 2016 will be included and studied. The investigators will request further clinical outcome data from 10 hospitals that provided the data for the International Post-PCI FFR registry before.

A standardized form of a spreadsheet, including standardized definitions of variables, was used to collect the individual patient data from the principal investigators of each qualified registry. Patient clinical, angiographic, and physiologic data at the time of index PCI were recorded and already collected at Seoul National University Hospital. As clinical outcome data of 2 years of follow-up after index PCI are already collected in the International Post-PCI FFR registry (NCT04684043), clinical outcome data after 2 years of index PCI will be collected by medical records until 2021.5 of each hospital. All submitted data were double-checked by a central monitoring team in Seoul National University Hospital. All patients' identifying numbers are anonymized as "Subject_No" and the investigators will request the patients' clinical outcome data using these anonymized identifying numbers of the patients. Also, the investigators will share collected data with collaborators, using these numbers.

ELIGIBILITY:
Inclusion Criteria:

- Patients who underwent PCI and post-PCI FFR measurements after angiographically successful stent implantation (residual stenosis < 20% by visual estimation)

Exclusion Criteria:

* Post-PCI TIMI (The Thrombolysis In Myocardial Infarction) flow of < 3
* Depressed left ventricular systolic function (ejection fraction < 30%)
* Culprit lesion for the acute coronary syndrome
* Graft vessel
* Collateral feeder
* In-stent stenosis
* Primary myocardial or valvular heart disease
* Patients with life expectancy < 2 years.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who were diagnosed as obstructive coronary artery disease and treated by DES and measured post PCI FFR after PCI.
Sampling Method: Non-Probability Sample
Enrollment: 2128 (Actual)
Dates: Start 2021-09-06 (Actual); Primary Completion 2022-05-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
The cumulative incidence (percent) of target vessel failure | 5 years
  Target vessel failure is a composite of cardiac death, target vessel myocardial infarction, and target vessel revascularization.
  The cumulative incidence will be calculated as Kaplan-Mier estimates at 5 years.

SECONDARY OUTCOMES:
The cumulative incidence (percent) of cardiac death or myocardial infarction | 5 years
  This outcome is a composite of cardiac death and target vessel myocardial infarction.
  The cumulative incidence will be calculated as Kaplan-Mier estimates at 5 years.
The cumulative incidence (percent) of target vessel myocardial infarction | 5 years
  Target vessel myocardial infarction is myocardial infarction that occurred in the target vessel in which post-PCI FFR was measured.
  The cumulative incidence will be calculated as Kaplan-Mier estimates at 5 years.
The cumulative incidence (percent) of target vessel revascularization | 5 years
  Target vessel revascularization is a revascularization event in the target vessel in which post-PCI FFR was measured.
  The cumulative incidence will be calculated as Kaplan-Mier estimates at 5 years.

OTHER OUTCOMES:
Cut-off value of post-PCI FFR | 5 years
  Define the best cut-off value for predicting future adverse events.
  The optimal cut-off value of post-PCI FFR for predicting outcomes was calculated based on maximizing the difference of log-rank statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Bon-Kwon Koo, MD, Study Chair — Seoul National University Hospital, Seoul, South Korea; Joon-Hyung Doh, MD, Principal Investigator — Inje University Ilsan Paik Hospital, Goyang, South Korea; Shao-Liang Chen, MD, Principal Investigator — Nanjing First Hospital, Nanjing Medical University, Nanjing, China; Tsunekazu Kakuta, MD, Principal Investigator — Tsuchiura Kyodo General Hospital; Hitoshi Matsuo, MD, Principal Investigator — Gifu Heart Center, Gifu, Japan; Chang-Wook Nam, MD, Principal Investigator — Keimyung University Dongsan Medical Center, Daegu, South Korea; Eun-Seok Shin, MD, Principal Investigator — Ulsan University Hospital, Ulsan, South Korea; Joo Myung Lee, MD, Principal Investigator — Samsung Medical Center; Akiko Matsuo, MD, Principal Investigator — Kyoto Second Red Cross Hospital, Kyoto, Japan; Hyun-Jong Lee, MD, Principal Investigator — Sejong General Hospital
Locations (1):
- Bon-Kwon Koo, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided
This issue has to be discussed with collaborators.

REFERENCES:
- [Background] Neumann FJ, Sousa-Uva M, Ahlsson A, Alfonso F, Banning AP, Benedetto U, Byrne RA, Collet JP, Falk V, Head SJ, Juni P, Kastrati A, Koller A, Kristensen SD, Niebauer J, Richter DJ, Seferovic PM, Sibbing D, Stefanini GG, Windecker S, Yadav R, Zembala MO; ESC Scientific Document Group. 2018 ESC/EACTS Guidelines on myocardial revascularization. Eur Heart J. 2019 Jan 7;40(2):87-165. doi: 10.1093/eurheartj/ehy394. No abstract available. PMID 30165437
- [Background] Fearon WF, Nishi T, De Bruyne B, Boothroyd DB, Barbato E, Tonino P, Juni P, Pijls NHJ, Hlatky MA; FAME 2 Trial Investigators. Clinical Outcomes and Cost-Effectiveness of Fractional Flow Reserve-Guided Percutaneous Coronary Intervention in Patients With Stable Coronary Artery Disease: Three-Year Follow-Up of the FAME 2 Trial (Fractional Flow Reserve Versus Angiography for Multivessel Evaluation). Circulation. 2018 Jan 30;137(5):480-487. doi: 10.1161/CIRCULATIONAHA.117.031907. Epub 2017 Nov 2. PMID 29097450
- [Background] Montalescot G, Brieger D, Dalby AJ, Park SJ, Mehran R. Duration of Dual Antiplatelet Therapy After Coronary Stenting: A Review of the Evidence. J Am Coll Cardiol. 2015 Aug 18;66(7):832-847. doi: 10.1016/j.jacc.2015.05.053. PMID 26271067
- [Background] Hwang D, Lee JM, Lee HJ, Kim SH, Nam CW, Hahn JY, Shin ES, Matsuo A, Tanaka N, Matsuo H, Lee SY, Doh JH, Koo BK. Influence of target vessel on prognostic relevance of fractional flow reserve after coronary stenting. EuroIntervention. 2019 Aug 29;15(5):457-464. doi: 10.4244/EIJ-D-18-00913. PMID 30561367
- [Background] Li SJ, Ge Z, Kan J, Zhang JJ, Ye F, Kwan TW, Santoso T, Yang S, Sheiban I, Qian XS, Tian NL, Rab TS, Tao L, Chen SL. Cutoff Value and Long-Term Prediction of Clinical Events by FFR Measured Immediately After Implantation of a Drug-Eluting Stent in Patients With Coronary Artery Disease: 1- to 3-Year Results From the DKCRUSH VII Registry Study. JACC Cardiovasc Interv. 2017 May 22;10(10):986-995. doi: 10.1016/j.jcin.2017.02.012. Epub 2017 Apr 26. PMID 28456699
- [Background] Rimac G, Fearon WF, De Bruyne B, Ikeno F, Matsuo H, Piroth Z, Costerousse O, Bertrand OF. Clinical value of post-percutaneous coronary intervention fractional flow reserve value: A systematic review and meta-analysis. Am Heart J. 2017 Jan;183:1-9. doi: 10.1016/j.ahj.2016.10.005. Epub 2016 Oct 11. PMID 27979031
- [Background] van Zandvoort LJC, Masdjedi K, Witberg K, Ligthart J, Tovar Forero MN, Diletti R, Lemmert ME, Wilschut J, de Jaegere PPT, Boersma E, Zijlstra F, Van Mieghem NM, Daemen J. Explanation of Postprocedural Fractional Flow Reserve Below 0.85. Circ Cardiovasc Interv. 2019 Feb;12(2):e007030. doi: 10.1161/CIRCINTERVENTIONS.118.007030. PMID 30732469
- [Background] Piroth Z, Toth GG, Tonino PAL, Barbato E, Aghlmandi S, Curzen N, Rioufol G, Pijls NHJ, Fearon WF, Juni P, De Bruyne B. Prognostic Value of Fractional Flow Reserve Measured Immediately After Drug-Eluting Stent Implantation. Circ Cardiovasc Interv. 2017 Aug;10(8):e005233. doi: 10.1161/CIRCINTERVENTIONS.116.005233. PMID 28790165
- [Background] Hwang D, Lee JM, Yang S, Chang M, Zhang J, Choi KH, Kim CH, Nam CW, Shin ES, Kwak JJ, Doh JH, Hoshino M, Hamaya R, Kanaji Y, Murai T, Zhang JJ, Ye F, Li X, Ge Z, Chen SL, Kakuta T, Koo BK. Role of Post-Stent Physiological Assessment in a Risk Prediction Model After Coronary Stent Implantation. JACC Cardiovasc Interv. 2020 Jul 27;13(14):1639-1650. doi: 10.1016/j.jcin.2020.04.041. PMID 32703590
- [Derived] Hwang D, Chung J, Yang S, Shin ES, Nam CW, Lee HJ, Matsuo H, Lee JM, Shiraishi J, Matsuo A, Doh JH, Chen SL, Kakuta T, Koo BK. Long-Term and Temporal Relationships Between Post-Stent Fractional Flow Reserve and Clinical Outcomes. JACC Cardiovasc Interv. 2025 Dec 8;18(23):2863-2874. doi: 10.1016/j.jcin.2025.09.034. PMID 41371783